CLINICAL TRIAL: NCT03524651
Title: Ferrous Acetyl-Aspartate Casein Formulation Evaluation Over Ferrous Sulfate in Iron Deficiency Anemia (ACCESS): A Double-Dummy Randomized Clinical Trial
Brief Title: Ferrous Acetyl-Aspartate Casein Formulation Evaluation Over Ferrous Sulfate in Iron Deficiency Anemia
Acronym: ACCESS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Uni-Pharma Kleon Tsetis Pharmaceutical Laboratories S.A. (Industry)
Collaborators: Attikon Hospital (Other); Amalia Fleming Prefecture General Hospital of Melissia (Unknown); G.Gennimatas General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Omalin-01/ACCESS
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Iron Deficiency Anemia
Keywords: Iron Deficiency Anemia; Fe-ASP; Casein; Iron protein acetyl aspartate; Restoration of decreased hemoglobin; Ferrous sulfate
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferrous sulfate

STUDY DESIGN:
Intervention Model Description: Double-dummy, blind, randomized, phase IV clinical trial
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ferrous sulfate (Active Comparator): Patients will take every day for 12 weeks two oral capsules of 150 mg ferrous sulfate delivering 47 mg of active elemental iron. Capsules should be taken orally either two hours before meal or two hours after meal. The same patients will take every day on exactly the same time for 12 weeks two placebo vials of 15 ml volume with excipients contained in the commercially available formulation Fe-Asp Omalin (Uni-Pharma SA).
  Interventions: Drug: Ferrous Sulfate
- Fe-ASP (Active Comparator): Patients will take every day for 12 weeks two oral placebo capsules. Capsules should be taken orally either two hours before meal or two hours after meal. The same patients will take every day on exactly the same time for 12 weeks two vials of 15 ml volume of the Fe-Asp preparation Omalin (Uni-Pharma SA) delivering 40 mg of elemental iron.
  Interventions: Drug: Fe-ASP

INTERVENTIONS:
Drug: Ferrous Sulfate — Blisters of 10 capsules containing 150 mg of ferrous sulfate.
  Other Names: Microfer
  Arms: Ferrous sulfate
Drug: Fe-ASP — Boxes of 10 vials of 15 ml containing 800 mg of Iron protein acetyl aspartate.
  Other Names: Omalin
  Arms: Fe-ASP
Drug: Ferrous Sulfate — Boxes of 10 vials of 15 ml containing inactive ingredients of Omalin.
  Other Names: Omalin placebo
  Arms: Ferrous sulfate
Drug: Fe-ASP — Blisters of 10 capsules containing inactive ingredients of Microfer.
  Other Names: Microfer placebo
  Arms: Fe-ASP

SUMMARY:
The scope of this study is to compare the efficacy of the new oral formulation of Fe-ASP to oral ferrous sulfate in patients with iron deficiency anemia (IDA) for the restoration of decreased circulating Hb. The improvement of symptoms of anemia, the restoration of biomarkers of iron deficiency into the normal range and the incidence of GI tract side effects are the study secondary endpoints.

DETAILED DESCRIPTION:
Anemia is a major problem in the general population affecting 5.6% in the United States. Iron deficiency is the most common cause of anemia. Although traditionally considered to be mainly a problem of underdeveloped countries, a recent epidemiological survey reported high incidence of iron deficiency anemia (IDA) in Europe in 2011. The incidence rate measured per 1,000 person-years was 8.18 in Belgium, 8.93 in Italy, 12.42 in Germany and 14.14 in Spain. Women were affected four-times more than men. The major causes of IDA are chronic blood loss, chronic disorders and excess needs.

The cornerstones of management of IDA are recognition and management of the cause of iron loss and efficient iron supplementation. Iron supplementation is usually done through oral formulations of iron. Three oral iron preparations are broadly used: ferrous sulfate, ferrous gluconate, and ferrous fumarate. The usual dosage is 325 mg (corresponding to 65 mg of elemental iron) two times a day. One major limitation with oral iron supplementation is GI side effects observed in almost 40% of cases. These are gastric discomfort, nausea, vomiting and constipation and they are caused due to the oxidation of ferrous irons in the stomach by acidic gastric fluid into insoluble salts.

A new formulation of iron conjugated to one N-acetyl-aspartate derivative of casein (Fe-ASP) has recently been developed. Due to the casein coating, it is anticipated that iron is converted to a smaller extent in the stomach into insoluble salts. In this way, more iron reaches the duodenum to become absorbed whereas GI side effects are less often. In parallel, animal studies have shown that casein itself primes the expression of enzymes that facilitate the absorption of iron across the duodenal mucosa.

This formulation is anticipated to be better tolerated for oral ingestion since iron is readily absorbed in the duodenum. The aim is to compare the efficacy of the new oral formulation of Fe-ASP to oral ferrous sulfate in patients with IDA for the restoration of decreased circulating Hb.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age equal to or more than 18 years
* Written informed consent provided by the patient
* Hb below 10g/dl, as defined by other trials
* Absolute red blood cell (RBC) count below 4.5 x 106/mm3 for men or 4.0 x 106/mm3 for women
* Mean corpuscular volume (MCV) of RBCs below 80 fl
* Mean corpuscular Hb (MCH) of RBCs below 27 pg
* Total ferritin below 30 ng/ml; this criterion is associated with sensitivity more than 99% for iron deficiency
* In the case of patients with anemia after GI tract hemorrhage, inclusion criteria 6 and 7 DO NOT apply for study inclusion.

Exclusion Criteria:

* Age below 18 years
* Denial to provide written informed consent
* Acute myelogenous or lymphoblastic leukemia
* Multiple myeloma
* Primary or secondary myelodysplastic syndrome
* Planning for start of chemotherapy within the first 30 days after inclusion in the trial
* Planning for start of radiotherapy within the first 30 days after inclusion in the trial
* Intake of erythropoietin
* Planning for start of erythropoietin within the first 30 days after inclusion in the trial
* Intake of chemotherapy the last six months
* Intake of radiotherapy the last six months
* Known hemochromatosis
* Known celiac disease
* Liver cirrhosis of Child-Pugh stage II or III
* Any active overt bleeding
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Comparative increase of baseline Hb | 4 weeks
  The primary study endpoint is the comparative increase of baseline Hb in each study group after the first 4 weeks of treatment. Since the daily amount of elemental iron delivered with the ferrous sulfate regimen is 94 mg and with the Fe-ASP regimen 80 mg, the increase of baseline Hb will be adjusted per mg of delivered elemental iron.

SECONDARY OUTCOMES:
Normalization of Hb | 4 weeks and 12 weeks
  Differences between the two groups of treatment in normalization of Hb; this is defined as Hb≥13 g/dl for mean and ≥12 g/dl for women.
Ferritin levels | 4 weeks and 12 weeks
  Differences between the two groups of treatment in ferritin levels.
Absolute reticulocyte count | 1 week, 4 weeks and 12 weeks
  Differences between the two groups of treatment in absolute reticulocyte count.
Absolute RBC count, Hb, MCV and MCH | 4 weeks and 12 weeks
  Differences between the two groups of treatment in absolute RBC count, Hb, MCV and MCH.
Fatigue symptoms of IDA | 4 weeks and 12 weeks
  Differences between the two groups of treatment in change of the fatigue symptoms of IDA.
Physical findings of IDA | 4 weeks and 12 weeks
  Differences between the two groups of treatment in change of physical findings of IDA.
Incidence of GI side effects | 4 weeks and 12 weeks
  Differences between the two groups of treatment in the incidence of GI side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Giamarellos-Bourboulis, MD, PhD, Principal Investigator — Attikon Hospital; Nikolaos Tsokos, MD, Principal Investigator — Amalia Fleming Prefecture General Hospital of Melissia; Georgios Adamis, MD, Principal Investigator — G.Gennimatas General Hospital
Locations (3):
- Greece (3):
  - General Hospital of Athens G. Gennimatas, Athens
  - Attikon University Hospital, Haidari/Athens
  - Amalia Fleming Prefecture General Hospital of Melissia, Melíssia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lazzari F, Carrara M. Overview of clinical trials in the treatment of iron deficiency with iron-acetyl-aspartylated casein. Clin Drug Investig. 2005;25(11):679-89. doi: 10.2165/00044011-200525110-00001. PMID 17532714